CLINICAL TRIAL: NCT03349060
Title: A PHASE 3 RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL GROUP, MULTI-CENTER STUDY TO EVALUATE THE EFFICACY AND SAFETY OF PF-04965842 MONOTHERAPY IN SUBJECTS AGED 12 YEARS AND OLDER, WITH MODERATE TO SEVERE ATOPIC DERMATITIS
Brief Title: Study to Evaluate Efficacy and Safety of PF-04965842 in Subjects Aged 12 Years And Older With Moderate to Severe Atopic Dermatitis
Acronym: JADE Mono-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B7451012; 2017-003651-29 (EudraCT Number); MONO-1 (Other: Alias Study Number); JADE MONO-1 (Other: Alias Study Number)
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Results first posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-11

CONDITIONS: Dermatitis, Atopic
Keywords: atopic dermatitis; atopic eczema; eczema; JAK; janus kinase
MeSH Terms: conditions — Dermatitis, Atopic; Eczema | interventions — abrocitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- PF-04965842 100 mg (Experimental)
  Interventions: Drug: PF-04965842 100 mg
- PF-04965842 200 mg (Experimental)
  Interventions: Drug: PF-04965842 200 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-04965842 100 mg — PF-04965842 100 mg, administered as two tablets to be taken orally once daily for 12 weeks
  Arms: PF-04965842 100 mg
Drug: PF-04965842 200 mg — PF-04965842 200 mg, administered as two tablets to be taken orally once daily for 12 weeks
  Arms: PF-04965842 200 mg
Drug: Placebo — Placebo, administered as two tablets to be taken orally once daily for 12 weeks
  Arms: Placebo

SUMMARY:
B7451012 is a Phase 3 study to evaluate PF-04965842 in patients aged 12 years and older with a minimum body weight of 40 kg who have moderate to severe atopic dermatitis. The efficacy and safety of two dosage strengths of PF-04965842, 100 mg and 200 mg taken orally once daily, will be evaluated relative to placebo over 12 weeks of study participation. Eligible patients will have an option to enter a long-term extension study after completing 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* 12 years of age or older with a minimum body weight of 40 kg
* Diagnosis of atopic dermatitis (AD) for at least 1 year and current status of moderate to severe disease (>= the following scores: BSA 10%, IGA 3, EASI 16, Pruritus NRS 4)
* Recent history of inadequate response or inability to tolerate topical AD treatments or require systemic treatments for AD control

Exclusion Criteria:

* Unwilling to discontinue current AD medications prior to the study or require treatment with prohibited medications during the study
* Prior treatment with JAK inhibitors
* Other active nonAD inflammatory skin diseases or conditions affecting skin
* Medical history including thrombocytopenia, coagulopathy or platelet dysfunction, Q wave interval abnormalities, current or history of certain infections, cancer, lymphoproliferative disorders and other medical conditions at the discretion of the investigator
* Pregnant or breastfeeding women, or women of childbearing potential who are unwilling to use contraception

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2017-12-07 (Actual); Primary Completion 2019-03-26 (Actual); Study Completion 2019-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (88):
- United States (29):
  - Clinical Research Center of Alabama, LLC, Birmingham, Alabama
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Rady Children's Hospital - San Diego/University of California, San Diego, San Diego, California
  - TCR Medical Corporation, San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - Florida Academic Centers Research and Education, LLC, Coral Gables, Florida
  - Olympian Clinical Research, Largo, Florida
  - Forward Clinical Trials, Inc., Tampa, Florida
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - NorthShore University HealthSystem Dermatology Clinical Trials Unit, Skokie, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Dawes Fretzin Dermatology Group, LLC, Indianapolis, Indiana
  - Tufts Medical Center, Boston, Massachusetts
  - Henry Ford Medical Center, New Center One, Detroit, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Medical University of South Carolina Investigational Drug Services, Charleston, South Carolina
  - MUSC SCTR Research Nexus Clinic and Laboratory, Charleston, South Carolina
  - Arlington Research Center, Inc., Arlington, Texas
  - The University of Texas Health Science Center Houston, Houston, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia
  - Pace Dermatology Associates, Lakewood, Washington
  - MultiCare Allenmore Hospital, Tacoma, Washington
  - MultiCare Institute for Research and Innovation, Tacoma, Washington
  - Pace Dermatology Associates, Tacoma, Washington
- Australia (10):
  - Australian Clinical Research Network (ACRN), Maroubra, New South Wales
  - Spectrum Medical Imaging, Maroubra, New South Wales
  - Queensland X-Ray, Upper Mount Gravatt, Queensland
  - Veracity Clinical Research Pty Ltd, Woolloongabba, Queensland
  - Emeritus Research, Camberwell, Victoria
  - Skin and Cancer Foundation Inc, Carlton, Victoria
  - Melbourne Radiology Clinic, East Melbourne, Victoria
  - Sinclair Dermatology, East Melbourne, Victoria
  - The Royal Children's Hospital, Parkville, Victoria
  - Bridge Road Imaging, Richmond, Victoria
- Canada (12):
  - Kirk Barber Research, Calgary, Alberta
  - Institute for Skin Advancement, Calgary, Alberta
  - Dr. Chih-ho Hong Medical Inc, Surrey, British Columbia
  - University of British Columbia Department of Dermatology and Skin Science, Vancouver, British Columbia
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - Lynderm Research Inc, Markham, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - The Centre for Dermatology, Richmond Hill, Ontario
  - York Dermatology Center, Richmond Hill, Ontario
  - Research Toronto, Toronto, Ontario
  - Innovaderm Research Inc., Montreal, Quebec
  - Diex Research Sherbrooke Inc., Sherbrooke, Quebec
- Czechia (8):
  - Lekarna Na Vaclavskem namesti, Kutná Hora
  - Kozni ambulance Kutna Hora, s.r.o., Kutná Hora
  - Lekarna Fakultni Nemocnice Ostrava, Ostrava - Poruba
  - Fakultni Nemocnice Ostrava, Kozni oddeleni, Ostrava - Poruba
  - Sanatorium profesora Arenbergera, Prague
  - Lekarna U sv. Ignace, Prague
  - Krajska zdravotni a.s.,Masarykova nemocnice o.z., Ústí nad Labem
  - Lekarna Masarykovy nemocnice v Usti nad Labem, o.z., Ústí nad Labem
- Germany (10):
  - Universitaetsklinikum Schleswig-Holstein/Campus Luebeck, Lübeck, Schleswig-Holstein
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Charité - Universitaetsmedizin Berlin, CCM, Berlin
  - ISA - Interdisciplinary Study Association GmbH, Berlin
  - Universitaetsklinikum Carl Gustav Carus der Technischen Universitaet Dresden, Dresden
  - Universitätsklinikum Erlangen, Hautklinik, Erlangen
  - Universitaetsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Ludwig-Maximilians-University Munich, Munich
  - Universitätsklinikum Münster, Münster
  - Klinische Forschung Schwerin GmbH, Schwerin
- Hungary (6):
  - Bács-Kiskun Megyei Kórház, Bőr-és nemibeteg Szakrendelés, Kecskemét, Bács-Kiskun county
  - Debreceni Egyetem Klinikai Kozpont Borgyogyaszati Klinika, Debrecen
  - Bacs-Kiskun Megyei Korhaz Kozponti Radiologiai Osztaly, Kecskemét
  - CRU Hungary Ltd., Miskolc
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Bor-,Nemikortani es Onkodermatologiai Klinika, Pécs
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
- Poland (8):
  - MULTIKLINIKA Salute Sp. z o.o., Katowice
  - Silmedic Sp. z o.o., Oddzial w Katowicach, Katowice
  - Centrum Medyczne Angelius Provita, Katowice
  - Pro Familia Altera Sp. z o.o., Katowice
  - NZOZ "DERMED" Centrum Medyczne Sp. z o.o. - Oddzial w Lodzi, Lodz
  - Dermoklinika Centrum Medyczne s.c., M. Kierstan, J. Narbutt, A. Lesiak, Lodz
  - Dermedic Jacek Zdybski, Ostrowiec Świętokrzyski
  - Wojskowy Instytut Medyczny, Klinika Dermatologiczna, Warsaw
- United Kingdom (5):
  - Derriford Hospital, Plymouth Hospitals NHS Trust, Plymouth, Devon
  - Royal Free London NHS Foundation Trust, London, Greater London
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, England
  - Sheffield Children's Hospital NHS Foundation Trust, Sheffield, South Yorkshire
  - The Dudley Group NHS Foundation Trust, Dudley

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Paller AS, Eichenfield LF, Irvine AD, Flohr C, Wollenberg A, Barbarot S, Bangert C, Spergel JM, Selfridge A, Biswas P, Fan H, Alderfer J, Watkins M, Koppensteiner H. Integrated Efficacy and Safety Analysis of Abrocitinib in Adolescents With Moderate-to-Severe Atopic Dermatitis. Allergy. 2025 Aug;80(8):2213-2224. doi: 10.1111/all.16512. Epub 2025 Mar 3. PMID 40028832
- [Derived] Silverberg JI, Thyssen JP, Lazariciu I, Myers DE, Guler E, Chovatiya R. Abrocitinib may improve itch and quality of life in patients with itch-dominant atopic dermatitis. Skin Health Dis. 2024 May 5;4(4):e382. doi: 10.1002/ski2.382. eCollection 2024 Aug. PMID 39104653
- [Derived] Armstrong AW, Alexis AF, Blauvelt A, Silverberg JI, Feeney C, Levenberg M, Chan G, Zhang F, Fostvedt L. Predicting Abrocitinib Efficacy at Week 12 Based on Clinical Response at Week 4: A Post Hoc Analysis of Four Randomized Studies in Moderate-to-Severe Atopic Dermatitis. Dermatol Ther (Heidelb). 2024 Jul;14(7):1849-1861. doi: 10.1007/s13555-024-01183-3. Epub 2024 Jun 19. PMID 38896380
- [Derived] Schmid-Grendelmeier P, Gooderham MJ, Hartmann K, Konstantinou GN, Fellmann M, Koulias C, Clibborn C, Biswas P, Brunner PM. Efficacy and safety of abrocitinib in patients with moderate-to-severe atopic dermatitis and comorbid allergies. Allergy. 2024 Jan;79(1):174-183. doi: 10.1111/all.15952. Epub 2023 Nov 21. PMID 37988255
- [Derived] Alexis AF, Silverberg JI, Rice ZP, Armstrong AW, Desai SR, Fonacier L, Kabashima K, Biswas P, Cella RR, Chan GL, Levenberg M. Abrocitinib efficacy and safety in moderate-to-severe atopic dermatitis by race, ethnicity, and Fitzpatrick skin type. Ann Allergy Asthma Immunol. 2024 Mar;132(3):383-389.e3. doi: 10.1016/j.anai.2023.11.002. Epub 2023 Nov 10. PMID 37949351
- [Derived] Blauvelt A, Boguniewicz M, Brunner PM, Luna PC, Biswas P, DiBonaventura M, Farooqui SA, Rojo R, Cameron MC. Abrocitinib monotherapy in Investigator's Global Assessment nonresponders: improvement in signs and symptoms of atopic dermatitis and quality of life. J Dermatolog Treat. 2022 Aug;33(5):2605-2613. doi: 10.1080/09546634.2022.2059053. Epub 2022 Jul 6. PMID 35763326
- [Derived] Stander S, Bhatia N, Gooderham MJ, Silverberg JI, Thyssen JP, Biswas P, DiBonaventura M, Romero W, Farooqui SA. High threshold efficacy responses in moderate-to-severe atopic dermatitis are associated with additional quality of life benefits: pooled analyses of abrocitinib monotherapy studies in adults and adolescents. J Eur Acad Dermatol Venereol. 2022 Aug;36(8):1308-1317. doi: 10.1111/jdv.18170. Epub 2022 May 6. PMID 35462428
- [Derived] Wojciechowski J, Malhotra BK, Wang X, Fostvedt L, Valdez H, Nicholas T. Population pharmacokinetic-pharmacodynamic modelling of platelet time-courses following administration of abrocitinib. Br J Clin Pharmacol. 2022 Aug;88(8):3856-3871. doi: 10.1111/bcp.15334. Epub 2022 Apr 11. PMID 35342978
- [Derived] Wojciechowski J, Malhotra BK, Wang X, Fostvedt L, Valdez H, Nicholas T. Population Pharmacokinetics of Abrocitinib in Healthy Individuals and Patients with Psoriasis or Atopic Dermatitis. Clin Pharmacokinet. 2022 May;61(5):709-723. doi: 10.1007/s40262-021-01104-z. Epub 2022 Jan 21. PMID 35061234
- [Derived] Cork MJ, McMichael A, Teng J, Valdez H, Rojo R, Chan G, Zhang F, Myers DE, DiBonaventura M. Impact of oral abrocitinib on signs, symptoms and quality of life among adolescents with moderate-to-severe atopic dermatitis: an analysis of patient-reported outcomes. J Eur Acad Dermatol Venereol. 2022 Mar;36(3):422-433. doi: 10.1111/jdv.17792. Epub 2021 Dec 4. PMID 34743361
- [Derived] Simpson EL, Silverberg JI, Nosbaum A, Winthrop KL, Guttman-Yassky E, Hoffmeister KM, Egeberg A, Valdez H, Zhang M, Farooqui SA, Romero W, Thorpe AJ, Rojo R, Johnson S. Integrated Safety Analysis of Abrocitinib for the Treatment of Moderate-to-Severe Atopic Dermatitis From the Phase II and Phase III Clinical Trial Program. Am J Clin Dermatol. 2021 Sep;22(5):693-707. doi: 10.1007/s40257-021-00618-3. Epub 2021 Aug 18. PMID 34406619
- [Derived] Silverberg JI, Thyssen JP, Simpson EL, Yosipovitch G, Stander S, Valdez H, Rojo R, Biswas P, Myers DE, Feeney C, DiBonaventura M. Impact of Oral Abrocitinib Monotherapy on Patient-Reported Symptoms and Quality of Life in Adolescents and Adults with Moderate-to-Severe Atopic Dermatitis: A Pooled Analysis of Patient-Reported Outcomes. Am J Clin Dermatol. 2021 Jul;22(4):541-554. doi: 10.1007/s40257-021-00604-9. Epub 2021 May 5. PMID 33954933
- [Derived] Simpson EL, Sinclair R, Forman S, Wollenberg A, Aschoff R, Cork M, Bieber T, Thyssen JP, Yosipovitch G, Flohr C, Magnolo N, Maari C, Feeney C, Biswas P, Tatulych S, Valdez H, Rojo R. Efficacy and safety of abrocitinib in adults and adolescents with moderate-to-severe atopic dermatitis (JADE MONO-1): a multicentre, double-blind, randomised, placebo-controlled, phase 3 trial. Lancet. 2020 Jul 25;396(10246):255-266. doi: 10.1016/S0140-6736(20)30732-7. PMID 32711801
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451012

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with age greater than or equal to (>=) 12 years with moderate to severe atopic dermatitis (AD) and a body weight of >=40 kilogram were enrolled in the study. Eligible participants had an option to enter into a long-term extension (LTE) study after completing 12 weeks of treatment in this study.
Pre-assignment Details: This study was conducted from 07-December-2017 to 26-March-2019 at 76 sites in 8 countries.
Groups:
- PF-04965842 100 mg: Participants were randomized to receive a tablet of PF-04965842 100 milligram (mg) and a tablet of matching placebo orally once daily for 12 weeks. Participants who discontinued early from treatment or who were not eligible for LTE study, were followed up to 4 weeks after last dose of study drug.
- PF-04965842 200 mg: Participants were randomized to receive PF-04965842 200 mg (2 tablets of 100 mg each) orally once daily for 12 weeks. Participants who discontinued early from treatment or who were not eligible for LTE study, were followed up to 4 weeks after last dose of study drug.
- Placebo: Participants were randomized to receive 2 tablets of placebo matched to PF-04965842 100 mg orally once daily for 12 weeks. Participants who discontinued early from treatment or who were not eligible for LTE study, were followed up to 4 weeks after last dose of study drug.
Period: Overall Study
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Started | 156 | 154 | 77
Completed | 135 | 137 | 61
Not Completed | 21 | 17 | 16
Not completed — Adverse Event | 9 | 9 | 7
Not completed — Lack of Efficacy | 1 | 0 | 2
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Protocol Violation | 2 | 2 | 1
Not completed — Withdrawal by Subject | 5 | 3 | 4
Not completed — Medication error,no linked adverse event | 0 | 0 | 1
Not completed — Withdrawal By Parent/Guardian | 0 | 1 | 0
Not completed — Other | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo | Total
Number analyzed (Participants) | 156 | 154 | 77 | 387
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.6 (15.4) | 33.0 (17.4) | 31.5 (14.4) | 32.5 (16.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 73 | 28 | 167
  Male | 90 | 81 | 49 | 220
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 4 | 6 | 20
  Not Hispanic or Latino | 144 | 149 | 71 | 364
  Unknown or Not Reported | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 4 | 1 | 6
  Asian | 26 | 26 | 6 | 58
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 15 | 11 | 6 | 32
  White | 113 | 104 | 62 | 279
  More than one race | 1 | 6 | 1 | 8
  Unknown or Not Reported | 0 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Investigator's Global Assessment (IGA) Response of Clear (0) or Almost Clear (1) and Greater Than or Equal to 2 Points Improvement From Baseline at Week 12
Description: IGA assesses severity of AD on a 5 point scale (0 to 4, higher scores indicate more severity). Scores: 0= clear, no inflammatory signs of AD; 1= almost clear, AD not fully cleared- light pink residual lesions (except post-inflammatory hyperpigmentation), just perceptible erythema, papulation/induration lichenification, excoriation, and no oozing/crusting; 2= mild AD with light red lesions, slight but definite erythema, papulation/induration, lichenification, excoriation and no oozing/crusting; 3= moderate AD with red lesions, moderate erythema, papulation/induration, lichenification, excoriation and slight oozing/crusting; 4= severe AD with deep dark red lesions, severe erythema, papulation/induration, lichenification, excoriation and moderate to severe oozing/crusting. Assessment excluded sole, palms and scalp.
Time Frame: Baseline, Week 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 76
percentage of participants | 23.7 | 43.8 | 7.9
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; The estimate and confidence interval (CI) for difference were calculated based on the weighted average of difference for each randomization stratum using the normal approximation of binomial proportions; Test type: Superiority; p = 0.0037, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 15.8, 95% CI 2-sided [6.8 to 24.8]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; The estimate and CI for difference were calculated based on the weighted average of difference for each randomization stratum using the normal approximation of binomial proportions; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 36.0, 95% CI 2-sided [26.2 to 45.7]

2. Primary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index (EASI) Response of >=75 Percent (%) Improvement From Baseline at Week 12
Description: EASI evaluates severity of participants' AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin)] and lower limbs [including buttocks]) on 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 156 | 153 | 76
percentage of participants | 39.7 | 62.7 | 11.8
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 27.9, 95% CI 2-sided [17.4 to 38.3]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Percentage = 51.0, 95% CI 2-sided [40.5 to 61.5]

3. Secondary Outcome: Percentage of Participants With at Least 4 Points Improvement From Baseline in the Numerical Rating Scale (NRS) for Severity of Pruritus at Week 2, 4, 8 and 12: Full Analysis Set (FAS)
Description: Participants were asked to assess their worst pruritus/itching due to AD over the past 24 hours on an NRS scale ranged from 0 (no itching) to 10 (worst possible itching), where higher scores indicated greater severity.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 147 | 147 | 74
percentage of participants
  Week 2 | 20.4 | 45.6 | 2.7
  Week 4 | 32.2 | 58.8 | 17.2
  Week 8 | 34.3 | 59.9 | 14.4
  Week 12 | 37.7 | 57.2 | 15.3
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; Week 2: Each complete imputed data set was analyzed using the Cochran-Mantel-Haenszel (CMH) risk difference method adjusting by randomization strata, separately for each week. Results from multiply imputed data sets were combined using Rubin's rules to obtain treatment difference, 95% CI and p-value; Test type: Superiority; p = 0.0004, Cochran-Mantel-Haenszel; Difference in Percentage = 18.0, 95% CI 2-sided [10.2 to 25.8]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; Week 2: Each complete imputed data set was analyzed using the CMH risk difference method adjusting by randomization strata, separately for each week. Results from multiply imputed data sets were combined using Rubin's rules to obtain treatment difference, 95% CI and p-value; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Percentage = 42.5, 95% CI 2-sided [33.6 to 51.4]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; Week 4: Each complete imputed data set was analyzed using the CMH risk difference method adjusting by randomization strata, separately for each week. Results from multiply imputed data sets were combined using Rubin's rules to obtain treatment difference, 95% CI and p-value; Test type: Superiority; p = 0.0251, Cochran-Mantel-Haenszel; Difference in Percentage = 15.0, 95% CI 2-sided [1.9 to 28.0]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Percentage = 41.1, 95% CI 2-sided [27.8 to 54.4]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; Week 8: Each complete imputed data set was analyzed using the CMH risk difference method adjusting by randomization strata, separately for each week. Results from multiply imputed data sets were combined using Rubin's rules to obtain treatment difference, 95% CI and p-value; Test type: Superiority; p = 0.0019, Cochran-Mantel-Haenszel; Difference in Percentage = 20.0, 95% CI 2-sided [7.4 to 32.7]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Percentage = 45.3, 95% CI 2-sided [32.7 to 57.8]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; Week 12: Each complete imputed data set was analyzed using the CMH risk difference method adjusting by randomization strata, separately for each week. Results from multiply imputed data sets were combined using Rubin's rules to obtain treatment difference, 95% CI and p-value; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel; Difference in Percentage = 22.5, 95% CI 2-sided [10.3 to 34.8]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Percentage = 41.7, 95% CI 2-sided [29.6 to 53.9]

4. Secondary Outcome: Percentage of Participants With at Least 4 Points Improvement From Baseline in the Numerical Rating Scale for Severity of Pruritus at Week 2, 4 and 12: Per Protocol Analysis Set (PPAS)
Description: as for outcome 3
Time Frame: Baseline, Week 2, 4, 12
Population: Per-protocol analysis set included all randomized participants who received at least 1 dose of study medication and who had no major protocol violations. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 127 | 126 | 54
percentage of participants
  Week 2 | 20.5 | 47.6 | 3.7
  Week 4 | 34.0 | 63.3 | 20.7
  Week 12 | 41.1 | 60.6 | 12.3
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.0055, Cochran-Mantel-Haenszel; Difference in Percentage = 16.3, 95% CI 2-sided [7.4 to 25.2]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Percentage = 43.3, 95% CI 2-sided [33.1 to 53.6]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p = 0.1138, Cochran-Mantel-Haenszel; Difference in Percentage = 12.5, 95% CI 2-sided [-3.0 to 28.0]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Percentage = 41.8, 95% CI 2-sided [26.2 to 57.4]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Percentage = 28.7, 95% CI 2-sided [15.3 to 42.1]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 3, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Percentage = 47.8, 95% CI 2-sided [34.6 to 61.1]

5. Secondary Outcome: Change From Baseline in Pruritus and Symptoms Assessment for Atopic Dermatitis (PSAAD) Total Score at Week 2, 4, 8 and 12: Full Analysis Set
Description: PSAAD is a daily participant reported symptom electronic diary. Participants rated their symptoms of AD over the past 24 hours, using 11 items (itchy skin, painful skin, dry skin, flaky skin, cracked skin, bumpy skin, red skin, discolored skin [lighter or darker], bleeding from skin, seeping or oozing fluid from skin [other than blood], and skin swelling). Participant had to think about all the areas of their body affected by their skin condition and chose the number that best described their experience for each of the 11 items, from 0 (no symptoms) to 10 (extreme symptoms), higher scores signified worse skin condition. Total PSAAD score = arithmetic mean of 11 items, 0 (no symptoms) to 10 (extreme symptoms), where higher score = worse skin condition.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 137 | 138 | 68
units on a scale
  Change at Week 2 | -1.5 [-1.7 to -1.2] | -2.1 [-2.3 to -1.8] | -0.5 [-0.8 to -0.1]
  Change at Week 4 | -1.8 [-2.1 to -1.5] | -3.0 [-3.2 to -2.7] | -0.7 [-1.1 to -0.3]
  Change at Week 8 | -2.2 [-2.5 to -1.8] | -3.1 [-3.5 to -2.8] | -1.2 [-1.7 to -0.7]
  Change at Week 12 | -2.2 [-2.6 to -1.9] | -3.2 [-3.6 to -2.8] | -1.1 [-1.7 to -0.6]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; Change at Week 2: MMRM contained fixed factors of treatment, week, treatment by week interaction, randomization strata (baseline disease severity and age category) and baseline value and used an unstructured covariance matrix; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in least squares (LS) mean = -1.0, 95% CI 2-sided [-1.4 to -0.6]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -1.6, 95% CI 2-sided [-2.0 to -1.2]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; Change at Week 4: MMRM contained fixed factors of treatment, week, treatment by week interaction, randomization strata (baseline disease severity and age category) and baseline value and used an unstructured covariance matrix; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -1.1, 95% CI 2-sided [-1.6 to -0.6]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -2.2, 95% CI 2-sided [-2.8 to -1.7]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; Change at Week 8: MMRM contained fixed factors of treatment, week, treatment by week interaction, randomization strata (baseline disease severity and age category) and baseline value and used an unstructured covariance matrix; Test type: Superiority; p = 0.0035, Mixed Models Analysis; Difference in LS mean = -0.9, 95% CI 2-sided [-1.5 to -0.3]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -1.9, 95% CI 2-sided [-2.5 to -1.3]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; Change at Week 12: MMRM contained fixed factors of treatment, week, treatment by week interaction, randomization strata (baseline disease severity and age category) and baseline value and used an unstructured covariance matrix; Test type: Superiority; p = 0.0010, Mixed Models Analysis; Difference in LS mean = -1.1, 95% CI 2-sided [-1.7 to -0.4]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -2.1, 95% CI 2-sided [-2.7 to -1.4]

6. Secondary Outcome: Change From Baseline in Pruritus and Symptoms Assessment for Atopic Dermatitis Total Score at Week 12: Per Protocol Analysis Set
Description: as for outcome 5
Time Frame: Baseline, Week 12
Population: as for outcome 4
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 115 | 117 | 50
units on a scale | -2.4 [-2.8 to -2.1] | -3.4 [-3.8 to -3.0] | -1.1 [-1.7 to -0.5]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; MMRM contained fixed factors of treatment, week, treatment by week interaction, randomization strata (baseline disease severity and age category) and baseline value and used an unstructured covariance matrix; Test type: Superiority; p = 0.0002, Mixed Models Analysis; Difference in LS mean = -1.3, 95% CI 2-sided [-2.0 to -0.6]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -2.3, 95% CI 2-sided [-3.0 to -1.6]

7. Secondary Outcome: Time to Achieve >=4 Points Improvement From Baseline in Numerical Rating Scale for Severity of Pruritus
Description: Participants were asked to assess their worst itching/pruritus due to AD over the past 24 hours on an NRS scale ranged from 0 (no itching) to 10 (worst itch imaginable), where higher scores indicated greater severity. 95% CI was based on the Brookmeyer and Crowley method.
Time Frame: Baseline up to Week 12
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 73 | 106 | 23
days | 84.0 [56.0 to NA] — Upper limit was not evaluable since very less events were observed. | 14.0 [11.0 to 29.0] | 92.0 [85.0 to NA] — Upper limit was not evaluable since very less events were observed.
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; Test type: Superiority; p = 0.0071, Log Rank — P-value was controlled by randomization strata
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; Test type: Superiority; p < 0.0001, Log Rank — P-value was controlled by randomization strata

8. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index Response of >=75% Improvement From Baseline at Week 2, 4 and 8
Description: as for outcome 2
Time Frame: Baseline, Week 2, 4, 8
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies the number of participants evaluable for the specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 155 | 154 | 77
percentage of participants
  Week 2 | 10.3 | 24.0 | 3.9
  Week 4: number analyzed (Participants) | 152 | 152 | 76
  Week 4 | 27.6 | 47.4 | 14.5
  Week 8: number analyzed (Participants) | 154 | 154 | 75
  Week 8 | 38.3 | 57.8 | 13.3
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; Week 2: The estimate and CI for difference were calculated based on the weighted average of difference for each randomization stratum using the normal approximation of binomial proportions; Test type: Superiority; p = 0.0869, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 6.5, 95% CI 2-sided [-0.3 to 13.3]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 20.3, 95% CI 2-sided [12.0 to 28.6]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; Week 4: The estimate and CI for difference were calculated based on the weighted average of difference for each randomization stratum using the normal approximation of binomial proportions; Test type: Superiority; p = 0.0259, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 13.1, 95% CI 2-sided [2.6 to 23.6]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 33.0, 95% CI 2-sided [21.7 to 44.2]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; Week 8: The estimate and CI for difference were calculated based on the weighted average of difference for each randomization stratum using the normal approximation of binomial proportions; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 25.0, 95% CI 2-sided [14.2 to 35.8]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 44.6, 95% CI 2-sided [33.6 to 55.6]

9. Secondary Outcome: Percentage of Participants Achieving Investigator's Global Assessment Response of Clear (0) or Almost Clear (1) and >=2 Points Improvement From Baseline at Week 2, 4 and 8
Description: as for outcome 1
Time Frame: Baseline, Week 2, 4, 8
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 155 | 154 | 77
percentage of participants
  Week 2 | 3.9 | 9.7 | 0
  Week 4: number analyzed (Participants) | 152 | 152 | 76
  Week 4 | 10.5 | 27.0 | 5.3
  Week 8: number analyzed (Participants) | 153 | 154 | 75
  Week 8 | 20.3 | 35.7 | 6.7
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0802, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 3.9, 95% CI 2-sided [-0.7 to 8.5]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0045, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 9.8, 95% CI 2-sided [4.0 to 15.7]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.1888, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 5.2, 95% CI 2-sided [-1.9 to 12.4]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 21.7, 95% CI 2-sided [13.0 to 30.5]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0071, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 13.8, 95% CI 2-sided [5.2 to 22.4]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 29.3, 95% CI 2-sided [19.8 to 38.7]

10. Secondary Outcome: Percentage of Participants Achieving Investigator's Global Assessment Response of Clear (0) at Week 2, 4, 8 and 12
Description: as for outcome 1
Time Frame: Week 2, 4, 8, 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication. Here, "Number Analyzed" signifies number of participants evaluable at the specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 156 | 154 | 77
percentage of participants
  Week 2: number analyzed (Participants) | 155 | 154 | 77
  Week 2 | 0 | 0 | 0
  Week 4: number analyzed (Participants) | 152 | 152 | 76
  Week 4 | 0 | 6.6 | 0
  Week 8: number analyzed (Participants) | 153 | 154 | 75
  Week 8 | 4.6 | 11.7 | 0
  Week 12: number analyzed (Participants) | 156 | 153 | 76
  Week 12 | 7.1 | 13.1 | 0
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; P-value could not be calculated since percentage of participants with event was 0; Difference in Percentage = 0.0, 95% CI 2-sided [-3.8 to 3.8]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; P-value could not be calculated since percentage of participants with event was 0; Difference in Percentage = 0.0, 95% CI 2-sided [-3.8 to 3.8]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; P-value could not be calculated since percentage of participants with event was 0; Difference in Percentage = 0.0, 95% CI 2-sided [-3.9 to 3.9]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.0234, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 6.5, 95% CI 2-sided [1.3 to 11.7]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0592, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 4.6, 95% CI 2-sided [-0.3 to 9.5]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0022, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 11.7, 95% CI 2-sided [5.5 to 17.9]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; Week 12: The estimate and CI for difference were calculated based on the weighted average of difference for each randomization stratum using the normal approximation of binomial proportions; Test type: Superiority; p = 0.0190, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 7.0, 95% CI 2-sided [1.7 to 12.3]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.0010, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 13.1, 95% CI 2-sided [6.7 to 19.4]

11. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index Response of >=50% Improvement From Baseline at Week 2, 4, 8 and 12
Description: as for outcome 2
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 156 | 154 | 77
percentage of participants
  Week 2: number analyzed (Participants) | 155 | 154 | 77
  Week 2 | 34.2 | 55.2 | 10.4
  Week 4: number analyzed (Participants) | 152 | 152 | 76
  Week 4 | 54.6 | 73.7 | 21.1
  Week 8: number analyzed (Participants) | 154 | 154 | 75
  Week 8 | 57.8 | 76.6 | 24.0
  Week 12: number analyzed (Participants) | 156 | 153 | 76
  Week 12 | 57.7 | 75.8 | 22.4
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 24.0, 95% CI 2-sided [13.9 to 34.1]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 45.1, 95% CI 2-sided [34.7 to 55.5]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 33.5, 95% CI 2-sided [21.6 to 45.4]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 52.7, 95% CI 2-sided [41.2 to 64.2]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 34.1, 95% CI 2-sided [21.9 to 46.3]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Difference in Percentage = 52.9, 95% CI 2-sided [41.3 to 64.6]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 35.3, 95% CI 2-sided [23.3 to 47.4]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 53.5, 95% CI 2-sided [42.0 to 65.0]

12. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index Response of >=90% Improvement From Baseline at Week 2, 4, 8 and 12
Description: as for outcome 2
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 156 | 154 | 77
percentage of participants
  Week 2: number analyzed (Participants) | 155 | 154 | 77
  Week 2 | 1.9 | 5.2 | 1.3
  Week 4: number analyzed (Participants) | 152 | 152 | 76
  Week 4 | 7.9 | 24.3 | 3.9
  Week 8: number analyzed (Participants) | 154 | 154 | 75
  Week 8 | 14.3 | 33.1 | 5.3
  Week 12: number analyzed (Participants) | 156 | 153 | 76
  Week 12 | 18.6 | 38.6 | 5.3
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.7285, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 0.6, 95% CI 2-sided [-3.9 to 5.2]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.1448, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 4.0, 95% CI 2-sided [-1.2 to 9.2]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.2576, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 3.9, 95% CI 2-sided [-2.6 to 10.5]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 20.4, 95% CI 2-sided [12.0 to 28.9]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0423, Cochran-Mantel-Haenszel; Difference in Percentage = 9.0, 95% CI 2-sided [1.3 to 16.8]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 28.0, 95% CI 2-sided [18.7 to 37.2]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.0066, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 13.3, 95% CI 2-sided [5.4 to 21.2]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 33.4, 95% CI 2-sided [24.3 to 42.5]

13. Secondary Outcome: Percentage of Participants Achieving Eczema Area and Severity Index Response of 100% Improvement From Baseline at Week 2, 4, 8 and 12
Description: as for outcome 2
Time Frame: Baseline, Week 2, 4, 8, 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication. Here, "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 156 | 154 | 77
percentage of participants
  Week 2: number analyzed (Participants) | 155 | 154 | 77
  Week 2 | 0 | 0 | 0
  Week 4: number analyzed (Participants) | 152 | 152 | 76
  Week 4 | 0 | 6.6 | 0
  Week 8: number analyzed (Participants) | 154 | 154 | 75
  Week 8 | 4.5 | 11.7 | 0
  Week 12: number analyzed (Participants) | 156 | 153 | 76
  Week 12 | 6.4 | 13.1 | 0
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; P-value could not be calculated since percentage of participants with events was 0; Difference in Percentage = 0.0, 95% CI 2-sided [-3.8 to 3.8]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; P-value could not be calculated since percentage of participants with events was 0; Difference in Percentage = 0.0, 95% CI 2-sided [-3.8 to 3.8]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; P-value could not be calculated since percentage of participants with events was 0; Difference in Percentage = 0.0, 95% CI 2-sided [-3.9 to 3.9]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.0234, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 6.5, 95% CI 2-sided [1.3 to 11.7]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0604, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 4.6, 95% CI 2-sided [-0.3 to 9.5]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0022, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 11.7, 95% CI 2-sided [5.5 to 17.9]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.0255, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 6.4, 95% CI 2-sided [1.2 to 11.6]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.0010, Cochran-Mantel-Haenszel; Difference in Percentage = 13.1, 95% CI 2-sided [6.7 to 19.4]

14. Secondary Outcome: Change From Baseline in Eczema Area and Severity Index Total Score at Week 2, 4, 8 and 12
Description: as for outcome 2
Time Frame: Baseline, Week 2, 4, 8, 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 156 | 154 | 77
units on a scale
  Change at Week 2 | -9.8 [-11.3 to -8.4] | -14.7 [-16.1 to -13.3] | -4.1 [-6.1 to -2.1]
  Change at Week 4 | -14.7 [-16.3 to -13.1] | -19.6 [-21.2 to -17.9] | -6.8 [-9.2 to -4.5]
  Change at Week 8 | -16.3 [-18.1 to -14.6] | -21.3 [-23.0 to -19.5] | -7.8 [-10.3 to -5.3]
  Change at Week 12 | -16.6 [-18.4 to -14.7] | -22.3 [-24.1 to -20.4] | -8.2 [-10.9 to -5.5]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -5.8, 95% CI 2-sided [-8.2 to -3.3]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -10.6, 95% CI 2-sided [-13.0 to -8.1]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -7.9, 95% CI 2-sided [-10.7 to -5.0]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -12.7, 95% CI 2-sided [-15.6 to -9.9]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -8.5, 95% CI 2-sided [-11.6 to -5.5]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -13.5, 95% CI 2-sided [-16.5 to -10.4]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -8.3, 95% CI 2-sided [-11.6 to -5.1]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -14.0, 95% CI 2-sided [-17.3 to -10.8]

15. Secondary Outcome: Change From Baseline in Percentage Body Surface Area at Week 2, 4, 8 and 12
Description: 4 body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's hand with fingers in a closed position) fitting in the affected area of a body region was estimated. Maximum number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint was equal to 10% for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. Percent BSA for a body region was calculated as = total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for an individual: arithmetic mean of % BSA of all 4 body regions, ranges from 0 to 100%, with higher values representing greater severity of AD.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage BSA
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 156 | 154 | 77
Percentage BSA
  Change at Week 2 | -11.8 [-14.3 to -9.4] | -18.8 [-21.3 to -16.4] | -4.0 [-7.6 to -0.5]
  Change at Week 4 | -20.2 [-23.0 to -17.4] | -27.0 [-29.8 to -24.2] | -8.5 [-12.5 to -4.5]
  Change at Week 8 | -23.2 [-26.3 to -20.2] | -31.5 [-34.6 to -28.5] | -8.9 [-13.3 to -4.5]
  Change at Week 12 | -25.1 [-28.3 to -22.0] | -33.4 [-36.6 to -30.3] | -11.4 [-16.0 to -6.8]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0004, Mixed Models Analysis; Difference in LS mean = -7.8, 95% CI 2-sided [-12.1 to -3.5]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -14.8, 95% CI 2-sided [-19.0 to -10.5]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -11.7, 95% CI 2-sided [-16.6 to -6.9]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -18.5, 95% CI 2-sided [-23.4 to -13.6]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -14.3, 95% CI 2-sided [-19.7 to -9.0]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -22.6, 95% CI 2-sided [-28.0 to -17.3]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -13.8, 95% CI 2-sided [-19.3 to -8.2]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -22.0, 95% CI 2-sided [-27.6 to -16.5]

16. Secondary Outcome: Percentage of Participants With Percentage Body Surface Area Less Than (<) 5% at Week 2, 4, 8 and 12
Description: 4 body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's hand with fingers in a closed position) fitting in the affected area of a body region was estimated. Maximum number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint was equal to 10% for head and neck, 5% for upper limb, 3.33% for trunk and 2.5% for lower limb. % BSA for a body region was calculated as = total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for an individual: arithmetic mean of % BSA of all 4 body regions, ranges from 0 to 100%, with higher values representing greater severity of AD.
Time Frame: Week 2, 4, 8, 12
Population: as for outcome 10
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 156 | 154 | 77
percentage of participants
  Week 2: number analyzed (Participants) | 155 | 154 | 77
  Week 2 | 2.6 | 5.2 | 1.3
  Week 4: number analyzed (Participants) | 152 | 152 | 76
  Week 4 | 8.6 | 27.6 | 3.9
  Week 8: number analyzed (Participants) | 154 | 154 | 75
  Week 8 | 16.2 | 33.1 | 6.7
  Week 12: number analyzed (Participants) | 156 | 153 | 76
  Week 12 | 21.2 | 38.6 | 5.3
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.5210, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 1.3, 95% CI 2-sided [-3.4 to 6.0]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.1416, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 4.0, 95% CI 2-sided [-1.3 to 9.3]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.2002, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 4.6, 95% CI 2-sided [-2.1 to 11.2]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 23.6, 95% CI 2-sided [15.1 to 32.2]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0434, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 9.6, 95% CI 2-sided [1.3 to 17.9]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 26.6, 95% CI 2-sided [17.1 to 36.2]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.0019, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 15.8, 95% CI 2-sided [7.5 to 24.0]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 33.3, 95% CI 2-sided [24.0 to 42.7]

17. Secondary Outcome: Percentage of Participants With Scoring Atopic Dermatitis (SCORAD) Response of >=50% Improvement From Baseline at Week 2, 4, 8 and 12
Description: SCORAD: scoring index for AD combining extent, severity, subjective symptoms. Extent (A): rule of 9 was used to calculate BSA affected by AD as a % of whole BSA for each body region- head and neck 9%; upper limbs 9% each; lower limbs 18% each; anterior trunk 18%; back 18%; 1% for genitals. The score for each body region was added to determine A (0-100). Severity (B): severity of each sign (erythema; edema; oozing; excoriation; skin thickening; dryness) was assessed as none=0, mild=1, moderate=2,severe=3. The severity scores were summed to give B (0-18). Subjective symptoms (C): pruritus and sleep, each of these 2 were scored by participant/caregiver using visual analogue scale (VAS) where "0" = no itch/no sleeplessness and "10" = the worst imaginable itch/sleeplessness, higher scores=worse symptoms. Scores for itch and sleeplessness were added to give 'C' (0-20). The SCORAD for an individual was calculated: A/5 + 7*B/2 + C; range from 0 to 103; higher values of SCORAD=worse outcome.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable at the specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 148 | 150 | 75
percentage of participants
  Week 2 | 14.9 | 34.0 | 4.0
  Week 4: number analyzed (Participants) | 145 | 148 | 70
  Week 4 | 34.5 | 50.7 | 12.9
  Week 8: number analyzed (Participants) | 146 | 148 | 72
  Week 8 | 36.3 | 54.1 | 12.5
  Week 12: number analyzed (Participants) | 145 | 146 | 73
  Week 12 | 36.6 | 56.8 | 16.4
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0151, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 10.8, 95% CI 2-sided [3.3 to 18.3]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 30.0, 95% CI 2-sided [21.0 to 39.0]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.0010, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 21.2, 95% CI 2-sided [10.2 to 32.3]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 37.9, 95% CI 2-sided [26.6 to 49.3]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0003, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 23.5, 95% CI 2-sided [12.6 to 34.3]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 41.7, 95% CI 2-sided [30.7 to 52.7]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.0026, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 19.6, 95% CI 2-sided [8.1 to 31.1]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 40.0, 95% CI 2-sided [28.3 to 51.7]

18. Secondary Outcome: Percentage of Participants With Scoring Atopic Dermatitis Response of >=75% Improvement From Baseline at Week 2, 4, 8 and 12
Description: SCORAD: scoring index for AD combining extent, severity, subjective symptoms. Extent (A): rule of 9 was used to calculate BSA affected by AD as a % of whole BSA for each body region- head and neck 9%; upper limbs 9% each; lower limbs 18% each; anterior trunk 18%; back 18%; 1% for genitals. The score for each body region was added to determine A (0-100). Severity (B): severity of each sign (erythema; edema; oozing; excoriation; skin thickening; dryness) was assessed as none (0), mild (1), moderate (2) or severe (3). The severity scores added to give B (0-18). Subjective symptoms (C): pruritus and sleep loss, each of these 2 were scored by participant/caregiver using VAS where "0" = no itch or no sleeplessness and "10" = the worst imaginable itch or sleeplessness, higher scores worse symptoms. Scores for itch and sleeplessness added to give 'C' (0-20). The SCORAD for an individual was calculated: A/5 + 7*B/2 + C; range from 0 to 103; higher values of SCORAD = worse outcome.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 148 | 150 | 75
percentage of participants
  Week 2 | 1.4 | 6.0 | 0
  Week 4: number analyzed (Participants) | 145 | 148 | 70
  Week 4 | 2.8 | 18.2 | 2.9
  Week 8: number analyzed (Participants) | 146 | 148 | 72
  Week 8 | 12.3 | 23.6 | 1.4
  Week 12: number analyzed (Participants) | 145 | 146 | 73
  Week 12 | 12.4 | 30.8 | 4.1
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.3151, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 1.3, 95% CI 2-sided [-2.9 to 5.6]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0292, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 6.0, 95% CI 2-sided [0.7 to 11.3]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.9402, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = -0.2, 95% CI 2-sided [-5.9 to 5.5]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.0019, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 15.3, 95% CI 2-sided [7.3 to 23.2]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0078, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 10.8, 95% CI 2-sided [4.2 to 17.4]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 22.2, 95% CI 2-sided [14.2 to 30.1]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.0528, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 8.2, 95% CI 2-sided [1.0 to 15.3]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 26.4, 95% CI 2-sided [17.6 to 35.3]

19. Secondary Outcome: Change From Baseline in Scoring Atopic Dermatitis: Visual Analogue Scale of Sleep Loss at Week 2, 4, 8 and 12
Description: as for outcome 18
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 154 | 153 | 77
units on a scale
  Change at Week 2 | -2.1 [-2.4 to -1.7] | -3.1 [-3.5 to -2.8] | -0.8 [-1.3 to -0.3]
  Change at Week 4 | -2.5 [-2.9 to -2.1] | -3.7 [-4.1 to -3.3] | -1.0 [-1.5 to -0.4]
  Change at Week 8 | -2.8 [-3.2 to -2.4] | -3.8 [-4.2 to -3.4] | -1.3 [-1.9 to -0.7]
  Change at Week 12 | -2.9 [-3.4 to -2.5] | -3.7 [-4.2 to -3.3] | -1.6 [-2.2 to -1.0]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -1.3, 95% CI 2-sided [-1.9 to -0.6]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -2.3, 95% CI 2-sided [-3.0 to -1.7]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -1.6, 95% CI 2-sided [-2.2 to -0.9]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -2.7, 95% CI 2-sided [-3.4 to -2.0]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -1.5, 95% CI 2-sided [-2.3 to -0.8]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -2.5, 95% CI 2-sided [-3.2 to -1.8]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.0005, Mixed Models Analysis; Difference in LS mean = -1.3, 95% CI 2-sided [-2.1 to -0.6]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -2.1, 95% CI 2-sided [-2.9 to -1.4]

20. Secondary Outcome: Change From Baseline in Scoring Atopic Dermatitis: Total Score at Week 2, 4, 8 and 12
Description: as for outcome 18
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 150 | 151 | 75
units on a scale
  Change at Week 2 | -16.4 [-18.7 to -14.2] | -24.4 [-26.7 to -22.2] | -5.5 [-8.7 to -2.4]
  Change at Week 4 | -23.1 [-25.8 to -20.4] | -32.6 [-35.3 to -29.9] | -10.5 [-14.4 to -6.7]
  Change at Week 8 | -26.0 [-29.1 to -23.0] | -33.7 [-36.7 to -30.7] | -11.7 [-16.0 to -7.4]
  Change at Week 12 | -27.0 [-30.2 to -23.7] | -35.5 [-38.7 to -32.3] | -13.6 [-18.3 to -9.0]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -10.9, 95% CI 2-sided [-14.8 to -7.0]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -18.9, 95% CI 2-sided [-22.7 to -15.1]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < .0001, Mixed Models Analysis; Difference in LS mean = -12.6, 95% CI 2-sided [-17.3 to -7.8]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < .0001, Mixed Models Analysis; Difference in LS mean = -22.1, 95% CI 2-sided [-26.8 to -17.3]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p < .0001, Mixed Models Analysis; Difference in LS mean = -14.3, 95% CI 2-sided [-19.5 to -9.0]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p < .0001, Mixed Models Analysis; Difference in LS mean = -22.0, 95% CI 2-sided [-27.2 to -16.7]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -13.3, 95% CI 2-sided [-19.0 to -7.7]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p < .0001, Mixed Models Analysis; Difference in LS mean = -21.9, 95% CI 2-sided [-27.5 to -16.3]

21. Secondary Outcome: Percentage of Participants Achieving >=1 Point Improvement From Baseline in Pruritus and Symptoms Assessment for Atopic Dermatitis at Week 2, 4, 8 and 12
Description: as for outcome 5
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 135 | 136 | 67
percentage of participants
  Week 2: number analyzed (Participants) | 133 | 135 | 67
  Week 2 | 51.1 | 68.9 | 28.4
  Week 4: number analyzed (Participants) | 134 | 132 | 67
  Week 4 | 62.7 | 77.3 | 44.8
  Week 8: number analyzed (Participants) | 133 | 136 | 67
  Week 8 | 60.9 | 69.1 | 44.8
  Week 12: number analyzed (Participants) | 132 | 128 | 66
  Week 12 | 61.4 | 70.3 | 40.9
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0028, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 22.3, 95% CI 2-sided [8.7 to 35.9]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 40.1, 95% CI 2-sided [27.1 to 53.2]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.0217, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 17.1, 95% CI 2-sided [2.8 to 31.4]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 32.2, 95% CI 2-sided [18.5 to 45.9]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0363, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 15.7, 95% CI 2-sided [1.4 to 30.0]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0011, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 23.7, 95% CI 2-sided [9.8 to 37.7]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.0080, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 20.1, 95% CI 2-sided [5.8 to 34.5]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 29.1, 95% CI 2-sided [15.0 to 43.3]

22. Secondary Outcome: Change From Baseline in Dermatology Life Quality Index (DLQI) at Week 2, 4, 8 and 12
Description: DLQI is a 10-item questionnaire that measures the impact of skin disease on participant's (aged above 17 years) quality of life over the last week. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicated more impact on quality of life. Scores from all 10 questions added up to give DLQI total score range from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of participants.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 121 | 119 | 60
units on a scale
  Change at Week 2 | -5.9 [-6.9 to -5.0] | -7.6 [-8.6 to -6.7] | -2.1 [-3.5 to -0.8]
  Change at Week 4 | -6.8 [-7.8 to -5.9] | -9.6 [-10.6 to -8.7] | -3.5 [-4.9 to -2.1]
  Change at Week 8 | -6.8 [-7.9 to -5.6] | -9.3 [-10.5 to -8.2] | -4.0 [-5.6 to -2.3]
  Change at Week 12 | -7.0 [-8.1 to -5.8] | -9.1 [-10.3 to -8.0] | -4.2 [-5.9 to -2.5]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -3.8, 95% CI 2-sided [-5.4 to -2.2]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -5.5, 95% CI 2-sided [-7.1 to -3.9]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.0001, Mixed Models Analysis; Difference in LS mean = -3.3, 95% CI 2-sided [-5.0 to -1.7]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < .0001, Mixed Models Analysis; Difference in LS mean = -6.1, 95% CI 2-sided [-7.8 to -4.5]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.0075, Mixed Models Analysis; Difference in LS mean = -2.8, 95% CI 2-sided [-4.8 to -0.7]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -5.3, 95% CI 2-sided [-7.4 to -3.3]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.0072, Mixed Models Analysis; Difference in LS mean = -2.8, 95% CI 2-sided [-4.8 to -0.8]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -4.9, 95% CI 2-sided [-6.9 to -2.9]

23. Secondary Outcome: Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) at Week 2, 4, 8 and 12
Description: CDLQI is a 10-item questionnaire that measures the impact of skin disease on adolescents (aged 12-17 years) quality of life over the last week. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. CDLQI total score was the sum of individual scores of question 1-10 and ranges from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of children.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 32 | 32 | 16
units on a scale
  Change at Week 2 | -4.5 [-5.8 to -3.2] | -5.8 [-7.1 to -4.5] | -3.3 [-5.1 to -1.4]
  Change at Week 4 | -5.3 [-6.7 to -4.0] | -8.2 [-9.5 to -6.8] | -1.8 [-3.8 to 0.2]
  Change at Week 8 | -5.2 [-6.9 to -3.6] | -7.5 [-9.2 to -5.9] | -3.1 [-5.6 to -0.6]
  Change at Week 12 | -6.4 [-7.9 to -5.0] | -7.5 [-8.9 to -6.0] | -3.9 [-6.1 to -1.7]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.2750, Mixed Models Analysis; Difference in LS mean = -1.3, 95% CI 2-sided [-3.5 to 1.0]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0280, Mixed Models Analysis; Difference in LS mean = -2.5, 95% CI 2-sided [-4.8 to -0.3]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.0051, Mixed Models Analysis; Difference in LS mean = -3.5, 95% CI 2-sided [-5.9 to -1.1]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -6.4, 95% CI 2-sided [-8.8 to -4.0]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.1706, Mixed Models Analysis; Difference in LS mean = -2.1, 95% CI 2-sided [-5.1 to 0.9]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.0048, Mixed Models Analysis; Difference in LS mean = -4.4, 95% CI 2-sided [-7.4 to -1.4]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.0629, Mixed Models Analysis; Difference in LS mean = -2.5, 95% CI 2-sided [-5.2 to 0.1]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.0100, Mixed Models Analysis; Difference in LS mean = -3.6, 95% CI 2-sided [-6.2 to -0.9]

24. Secondary Outcome: Percentage of Participants With Baseline Dermatology Life Quality Index Score >=2 and Achieving <2 DLQI Score at Week 2, 4, 8 and 12
Description: as for outcome 22
Time Frame: Baseline, Week 2, 4, 8, 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 120 | 119 | 59
percentage of participants
  Week 2 | 10.0 | 23.5 | 3.4
  Week 4: number analyzed (Participants) | 118 | 117 | 59
  Week 4 | 15.3 | 32.5 | 8.5
  Week 8: number analyzed (Participants) | 118 | 119 | 57
  Week 8 | 17.8 | 35.3 | 8.8
  Week 12: number analyzed (Participants) | 119 | 119 | 58
  Week 12 | 20.2 | 31.9 | 12.1
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.1238, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 6.6, 95% CI 2-sided [-0.7 to 13.9]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0008, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 20.1, 95% CI 2-sided [11.0 to 29.2]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.2091, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 6.8, 95% CI 2-sided [-2.8 to 16.4]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.0005, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 24.0, 95% CI 2-sided [12.9 to 35.0]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.1161, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 9.1, 95% CI 2-sided [-0.9 to 19.1]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 26.5, 95% CI 2-sided [15.3 to 37.7]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.1837, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 8.1, 95% CI 2-sided [-2.8 to 19.1]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.0046, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 19.8, 95% CI 2-sided [8.1 to 31.6]

25. Secondary Outcome: Percentage of Participants With Baseline Children's Dermatology Life Quality Index Score >=2 and Achieving <2 CDLQI Score at Week 2, 4, 8 and 12
Description: as for outcome 23
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 24
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 31 | 31 | 16
percentage of participants
  Week 2 | 3.2 | 0 | 0
  Week 4: number analyzed (Participants) | 30 | 31 | 15
  Week 4 | 13.3 | 9.7 | 0
  Week 8: number analyzed (Participants) | 31 | 31 | 14
  Week 8 | 12.9 | 12.9 | 7.1
  Week 12: number analyzed (Participants) | 31 | 31 | 15
  Week 12 | 19.4 | 9.7 | 0
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.4795, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 3.2, 95% CI 2-sided [-10.3 to 16.6]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; P-value could not be calculated since percentage of participants with events was 0; Difference in Percentage = 0.0, 95% CI 2-sided [-12.7 to 12.7]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.1452, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 13.3, 95% CI 2-sided [-3.6 to 30.3]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.2232, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 9.7, 95% CI 2-sided [-6.1 to 25.4]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.5707, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 5.8, 95% CI 2-sided [-13.7 to 25.4]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.5777, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 5.8, 95% CI 2-sided [-13.6 to 25.1]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.0744, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 19.3, 95% CI 2-sided [1.0 to 37.5]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.2232, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 9.7, 95% CI 2-sided [-6.1 to 25.4]

26. Secondary Outcome: Percentage of Participants With Baseline Dermatology Life Quality Index Score >=4 and Achieving >=4 Point Improvement From Baseline in DLQI Score at Week 2, 4, 8 and 12
Description: as for outcome 22
Time Frame: Baseline, Week 2, 4, 8, 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" signifies participant who were evaluable for this measure and "Number Analyzed" signifies number of participants evaluable at specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 117 | 117 | 56
percentage of participants
  Week 2 | 67.5 | 71.8 | 35.7
  Week 4: number analyzed (Participants) | 115 | 115 | 56
  Week 4 | 72.2 | 85.2 | 51.8
  Week 8: number analyzed (Participants) | 116 | 117 | 54
  Week 8 | 64.7 | 82.1 | 48.1
  Week 12: number analyzed (Participants) | 116 | 117 | 55
  Week 12 | 67.2 | 72.6 | 43.6
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 31.6, 95% CI 2-sided [17.2 to 46.0]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 35.7, 95% CI 2-sided [21.5 to 49.9]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.0090, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 20.4, 95% CI 2-sided [5.2 to 35.6]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 33.3, 95% CI 2-sided [19.0 to 47.7]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0421, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 16.5, 95% CI 2-sided [0.6 to 32.4]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 33.8, 95% CI 2-sided [18.9 to 48.8]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.0035, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 23.5, 95% CI 2-sided [8.2 to 38.8]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 28.8, 95% CI 2-sided [13.8 to 43.9]

27. Secondary Outcome: Percentage of Participants With Baseline Children's Dermatology Life Quality Index Score >=2.5 and Achieving >=2.5 Point Improvement From Baseline in CDLQI Score at Week 2, 4, 8 and 12
Description: as for outcome 23
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 30 | 31 | 16
percentage of participants
  Week 2 | 73.3 | 74.2 | 56.3
  Week 4: number analyzed (Participants) | 29 | 31 | 15
  Week 4 | 69.0 | 83.9 | 40.0
  Week 8: number analyzed (Participants) | 30 | 31 | 14
  Week 8 | 66.7 | 77.4 | 35.7
  Week 12: number analyzed (Participants) | 30 | 31 | 15
  Week 12 | 73.3 | 83.9 | 53.3
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.2497, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 17.1, 95% CI 2-sided [-9.1 to 43.2]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.2371, Cochran-Mantel-Haenszel; Difference in Percentage = 17.1, 95% CI 2-sided [-9.0 to 43.3]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.0697, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 28.8, 95% CI 2-sided [-0.8 to 58.3]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.0030, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 43.9, 95% CI 2-sided [16.2 to 71.7]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0583, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 31.0, 95% CI 2-sided [2.0 to 59.9]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0085, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 41.2, 95% CI 2-sided [13.2 to 69.1]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.1948, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 19.3, 95% CI 2-sided [-9.8 to 48.5]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.0296, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 30.6, 95% CI 2-sided [2.8 to 58.5]

28. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS): Depression Subscale at Week 2, 4, 8 and 12
Description: HADS: participant rated 14-item questionnaire. HADS consisted of 2 subscales: HADS-anxiety scale (HADS-A) and HADS-depression scale (HADS-D), both of these subscales comprised of 7 items each. Each item was rated on a 4-point scale, score range from 0 to 3, where higher scores indicates more anxiety/depression symptoms. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks). HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). HADS-D: sum of all 7 items resulted in score range of 0 (no presence of depression) to 21 (severe feeling of depression); higher score indicating greater severity of depression symptoms.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 152 | 152 | 76
units on a scale
  Change at Week 2 | -0.7 [-1.0 to -0.3] | -1.3 [-1.6 to -0.9] | -0.2 [-0.7 to 0.3]
  Change at Week 4 | -1.1 [-1.6 to -0.7] | -1.7 [-2.1 to -1.3] | 0.1 [-0.5 to 0.7]
  Change at Week 8 | -1.0 [-1.4 to -0.6] | -2.0 [-2.4 to -1.6] | -0.3 [-0.9 to 0.3]
  Change at Week 12 | -1.4 [-1.8 to -0.9] | -1.8 [-2.2 to -1.4] | -0.2 [-0.8 to 0.4]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.1718, Mixed Models Analysis; Difference in LS mean = -0.5, 95% CI 2-sided [-1.1 to 0.2]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0018, Mixed Models Analysis; Difference in LS mean = -1.1, 95% CI 2-sided [-1.7 to -0.4]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.0005, Mixed Models Analysis; Difference in LS mean = -1.3, 95% CI 2-sided [-2.0 to -0.6]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -1.8, 95% CI 2-sided [-2.5 to -1.1]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.0476, Mixed Models Analysis; Difference in LS mean = -0.7, 95% CI 2-sided [-1.5 to -0.0]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -1.7, 95% CI 2-sided [-2.4 to -1.0]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.0028, Mixed Models Analysis; Difference in LS mean = -1.1, 95% CI 2-sided [-1.9 to -0.4]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -1.6, 95% CI 2-sided [-2.3 to -0.9]

29. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale: Anxiety Subscale at Week 2, 4, 8 and 12
Description: HADS: participant rated 14-item questionnaire. HADS consisted of 2 subscales: HADS-anxiety scale (HADS-A) and HADS-depression scale (HADS-D), both of these subscales comprised of 7 items each. Each item was rated on a 4-point scale, score range from 0 to 3, where higher scores indicates more anxiety/depression symptoms. HADS-A assesses state of generalized anxiety (anxious mood, restlessness, anxious thoughts, panic attacks). HADS-D assesses state of lost interest and diminished pleasure response (lowering of hedonic tone). HADS-A: sum of all 7 items resulted in score range of 0 (no presence of anxiety) to 21 (severe feeling of anxiety); higher score indicating greater severity of anxiety.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 152 | 152 | 76
units on a scale
  Change at Week 2 | -1.1 [-1.5 to -0.7] | -1.7 [-2.0 to -1.3] | -0.9 [-1.5 to -0.4]
  Change at Week 4 | -1.4 [-1.9 to -1.0] | -2.2 [-2.6 to -1.8] | -1.0 [-1.6 to -0.4]
  Change at Week 8 | -1.5 [-1.9 to -1.0] | -2.3 [-2.7 to -1.8] | -1.0 [-1.7 to -0.4]
  Change at Week 12 | -1.6 [-2.0 to -1.1] | -2.1 [-2.5 to -1.6] | -1.0 [-1.7 to -0.4]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.6134, Mixed Models Analysis; Difference in LS mean = -0.2, 95% CI 2-sided [-0.9 to 0.5]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0422, Mixed Models Analysis; Difference in LS mean = -0.7, 95% CI 2-sided [-1.4 to -0.0]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.2050, Mixed Models Analysis; Difference in LS mean = -0.5, 95% CI 2-sided [-1.2 to 0.3]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.0012, Mixed Models Analysis; Difference in LS mean = -1.2, 95% CI 2-sided [-1.9 to -0.5]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.2657, Mixed Models Analysis; Difference in LS mean = -0.4, 95% CI 2-sided [-1.2 to 0.3]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.0019, Mixed Models Analysis; Difference in LS mean = -1.2, 95% CI 2-sided [-2.0 to -0.5]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.1675, Mixed Models Analysis; Difference in LS mean = -0.5, 95% CI 2-sided [-1.3 to 0.2]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.0085, Mixed Models Analysis; Difference in LS mean = -1.0, 95% CI 2-sided [-1.8 to -0.3]

30. Secondary Outcome: Percentage of Participants With >=8 Points at Baseline and Achieving Score of <8 Points in Hospital Anxiety and Depression Scale: Anxiety Subscale at Week 2, 4, 8 and 12
Description: as for outcome 29
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 33 | 34 | 18
percentage of participants
  Week 2 | 48.5 | 64.7 | 38.9
  Week 4: number analyzed (Participants) | 32 | 33 | 18
  Week 4 | 50.0 | 54.5 | 55.6
  Week 8 | 42.4 | 58.8 | 22.2
  Week 12: number analyzed (Participants) | 33 | 33 | 18
  Week 12 | 39.4 | 48.5 | 38.9
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.5539, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 8.8, 95% CI 2-sided [-19.6 to 37.2]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0561, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 27.9, 95% CI 2-sided [0.8 to 55.1]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.7460, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = -4.9, 95% CI 2-sided [-33.4 to 23.7]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 1.0000, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = -0.0, 95% CI 2-sided [-28.3 to 28.3]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.1474, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 20.8, 95% CI 2-sided [-4.5 to 46.2]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0123, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 37.3, 95% CI 2-sided [12.1 to 62.5]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.9760, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = -0.4, 95% CI 2-sided [-28.5 to 27.6]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.5965, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 7.8, 95% CI 2-sided [-20.4 to 36.1]

31. Secondary Outcome: Percentage of Participants With >=8 Points at Baseline and Achieving Score of <8 Points in Hospital Anxiety and Depression Scale: Depression Subscale at Week 2, 4, 8 and 12
Description: as for outcome 28
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 22 | 20 | 9
percentage of participants
  Week 2 | 45.5 | 60.0 | 22.2
  Week 4: number analyzed (Participants) | 22 | 19 | 9
  Week 4 | 68.2 | 68.4 | 55.6
  Week 8: number analyzed (Participants) | 21 | 20 | 9
  Week 8 | 57.1 | 70.0 | 66.7
  Week 12 | 50.0 | 75.0 | 33.3
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.2278, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 24.0, 95% CI 2-sided [-9.9 to 58.0]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0996, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 35.2, 95% CI 2-sided [-2.0 to 72.4]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.4449, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 14.5, 95% CI 2-sided [-21.6 to 50.6]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.4139, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 16.9, 95% CI 2-sided [-21.6 to 55.5]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.7290, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = -6.7, 95% CI 2-sided [-40.7 to 27.4]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.6585, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 8.7, 95% CI 2-sided [-27.3 to 44.6]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.3638, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 18.2, 95% CI 2-sided [-18.7 to 55.1]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.0550, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 40.5, 95% CI 2-sided [2.4 to 78.5]

32. Secondary Outcome: Percentage of Participants With >=11 Points at Baseline and Achieving Score of <11 Points in Hospital Anxiety and Depression Scale: Anxiety Subscale at Week 2, 4, 8 and 12
Description: as for outcome 29
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 17
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 16 | 13 | 8
percentage of participants
  Week 2 | 56.3 | 46.2 | 75.0
  Week 4: number analyzed (Participants) | 16 | 12 | 8
  Week 4 | 56.3 | 58.3 | 75.0
  Week 8 | 56.3 | 53.8 | 75.0
  Week 12 | 43.8 | 46.2 | 37.5
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.4036, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = -18.8, 95% CI 2-sided [-58.4 to 20.9]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.1580, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = -35.3, 95% CI 2-sided [-75.9 to 5.3]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.5140, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = -14.2, 95% CI 2-sided [-53.5 to 25.1]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.4149, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = -19.8, 95% CI 2-sided [-63.3 to 23.7]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.4036, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = -18.8, 95% CI 2-sided [-58.4 to 20.9]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.2092, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = -30.7, 95% CI 2-sided [-70.9 to 9.6]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.5982, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 11.9, 95% CI 2-sided [-29.1 to 53.0]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.8647, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 4.2, 95% CI 2-sided [-36.3 to 44.7]

33. Secondary Outcome: Percentage of Participants With >=11 Points at Baseline and Achieving Score of <11 Points in Hospital Anxiety and Depression Scale: Depression Subscale at Week 2, 4, 8 and 12
Description: as for outcome 28
Time Frame: Baseline, Week 2, 4, 8, 12
Population: Full analysis set included all randomized participants who received at least 1 dose of study medication. Here, "Overall Number of Participants Analyzed" participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 5 | 8 | 3
percentage of participants
  Week 2 | 20.0 | 75.0 | 100.0
  Week 4 | 60.0 | 75.0 | 66.7
  Week 8 | 40.0 | 75.0 | 66.7
  Week 12 | 40.0 | 75.0 | 66.7
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0546, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = -78.6, 95% CI 2-sided [-117.5 to -39.6]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.3573, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = -27.9, 95% CI 2-sided [-62.5 to 6.7]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.9219, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = -3.6, 95% CI 2-sided [-55.6 to 48.5]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.3173, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 24.6, 95% CI 2-sided [-14.4 to 63.6]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.5408, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = -25.0, 95% CI 2-sided [-77.0 to 27.0]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.3173, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 24.6, 95% CI 2-sided [-14.4 to 63.6]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs PF-04965842 200 mg; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.5408, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = -25.0, 95% CI 2-sided [-77.0 to 27.0]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.3173, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 24.6, 95% CI 2-sided [-14.4 to 63.6]

34. Secondary Outcome: Change From Baseline in Patient-Oriented Eczema Measure (POEM) at Week 2, 4, 8 and 12
Description: POEM is a 7-item participant reported outcome (PRO) measure used to assess the impact of AD (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) over the past week. Each item is scored as "no days (0)", "1-2 days (1)", "3-4 days (2)", "5-6 days (3)" and "every day (4)". The score ranges from 0 to 28, where higher score indicated greater severity.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 153 | 153 | 77
units on a scale
  Change at Week 2 | -4.6 [-5.5 to -3.7] | -8.1 [-9.0 to -7.2] | -1.8 [-3.1 to -0.5]
  Change at Week 4 | -6.2 [-7.2 to -5.1] | -10.8 [-11.8 to -9.8] | -2.4 [-3.9 to -0.9]
  Change at Week 8 | -6.1 [-7.3 to -4.9] | -10.6 [-11.8 to -9.5] | -3.4 [-5.1 to -1.7]
  Change at Week 12 | -6.8 [-8.0 to -5.6] | -10.6 [-11.8 to -9.4] | -3.7 [-5.5 to -1.9]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0006, Mixed Models Analysis; Difference in LS mean = -2.8, 95% CI 2-sided [-4.4 to -1.2]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -6.3, 95% CI 2-sided [-7.9 to -4.7]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -3.8, 95% CI 2-sided [-5.6 to -2.0]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -8.4, 95% CI 2-sided [-10.2 to -6.6]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.0096, Mixed Models Analysis; Difference in LS mean = -2.7, 95% CI 2-sided [-4.7 to -0.7]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -7.2, 95% CI 2-sided [-9.3 to -5.2]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.0049, Mixed Models Analysis; Difference in LS mean = -3.1, 95% CI 2-sided [-5.2 to -0.9]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -6.9, 95% CI 2-sided [-9.0 to -4.7]

35. Secondary Outcome: Change From Baseline in Patient Global Assessment (PtGA) at Week 2, 4, 8 and 12
Description: Participant responded to "Overall, how would you describe your Atopic Dermatitis right now?" on a scale: 0= clear; 1= almost clear; 2= mild; 3= moderate; and 4= severe. Higher scores indicated more severity.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 154 | 153 | 77
units on a scale
  Change at Week 2 | -0.6 [-0.8 to -0.5] | -1.1 [-1.2 to -0.9] | -0.3 [-0.5 to -0.1]
  Change at Week 4 | -0.8 [-1.0 to -0.7] | -1.3 [-1.5 to -1.2] | -0.4 [-0.6 to -0.1]
  Change at Week 8 | -1.0 [-1.1 to -0.8] | -1.4 [-1.6 to -1.2] | -0.5 [-0.7 to -0.2]
  Change at Week 12 | -1.0 [-1.2 to -0.9] | -1.5 [-1.7 to -1.3] | -0.5 [-0.8 to -0.3]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0020, Mixed Models Analysis; Difference in LS mean = -0.4, 95% CI 2-sided [-0.6 to -0.1]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -0.8, 95% CI 2-sided [-1.0 to -0.6]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.0011, Mixed Models Analysis; Difference in LS mean = -0.5, 95% CI 2-sided [-0.7 to -0.2]
Statistical Analysis 4: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -1.0, 95% CI 2-sided [-1.2 to -0.7]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.0020, Mixed Models Analysis; Difference in LS mean = -0.5, 95% CI 2-sided [-0.8 to -0.2]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -0.9, 95% CI 2-sided [-1.2 to -0.6]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.0014, Mixed Models Analysis; Difference in LS mean = -0.5, 95% CI 2-sided [-0.8 to -0.2]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = -0.9, 95% CI 2-sided [-1.3 to -0.6]

36. Secondary Outcome: Percentage of Participants Achieving 'Clear' or 'Almost Clear' and >=2 Points Improvement From Baseline in Patient Global Assessment (PtGA) at Week 2, 4, 8 and 12
Description: as for outcome 35
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 8
Measure: Number; unit: percentage of participants
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 153 | 151 | 75
percentage of participants
  Week 2 | 7.2 | 19.2 | 1.3
  Week 4: number analyzed (Participants) | 151 | 149 | 74
  Week 4 | 14.6 | 31.5 | 5.4
  Week 8: number analyzed (Participants) | 151 | 151 | 71
  Week 8 | 17.2 | 34.4 | 8.5
  Week 12: number analyzed (Participants) | 152 | 150 | 73
  Week 12 | 21.1 | 36.0 | 6.8
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0575, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 6.0, 95% CI 2-sided [0.3 to 11.7]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 1]; Test type: Superiority; p = 0.0002, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 18.1, 95% CI 2-sided [10.7 to 25.5]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p = 0.0411, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 9.2, 95% CI 2-sided [1.3 to 17.1]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 3]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 26.2, 95% CI 2-sided [16.9 to 35.5]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p = 0.0781, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 8.9, 95% CI 2-sided [-0.1 to 18.0]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 8, analysis 5]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 26.2, 95% CI 2-sided [16.2 to 36.3]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p = 0.0075, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 14.2, 95% CI 2-sided [5.3 to 23.2]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 10, analysis 7]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — P-value was adjusted by randomization strata (baseline disease severity and age category); Difference in Percentage = 29.3, 95% CI 2-sided [19.6 to 38.9]

37. Secondary Outcome: Change From Baseline in EuroQol Quality of Life 5-Dimension 5-Level Scale (EQ-5D-5L): Index Value at Week 2, 4, 8 and 12
Description: EQ-5D-5L: standardized participant (aged >17 years) completed questionnaire consisted of 2 components: a health state profile and an optional VAS. EQ-5D health state profile had 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. Responses to 5 dimensions comprised a health state/a single utility index value. E.g. if a participant responded "no problems" for each 5 dimensions, then health state was coded as "11111" with a predefined index value to it. Every health state (coded as combination of responses on each of 5 dimensions) had a unique predefined utility index value assigned to it, by EuroQol. US value sets (with all possible health states) was used for adults in the study, range from 1 to -0.109. Higher (positive) scores = better health state.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 121 | 119 | 60
units on a scale
  Change at Week 2 | 0.049 [0.030 to 0.068] | 0.084 [0.065 to 0.103] | 0.016 [-0.011 to 0.043]
  Change at Week 4 | 0.062 [0.041 to 0.084] | 0.092 [0.070 to 0.114] | 0.037 [0.007 to 0.067]
  Change at Week 8 | 0.053 [0.029 to 0.077] | 0.097 [0.074 to 0.121] | 0.005 [-0.029 to 0.039]
  Change at Week 12 | 0.058 [0.034 to 0.083] | 0.078 [0.054 to 0.103] | 0.014 [-0.021 to 0.050]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0453, Mixed Models Analysis; Difference in LS mean = 0.034, 95% CI 2-sided [0.001 to 0.066]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = 0.068, 95% CI 2-sided [0.036 to 0.101]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.1821, Mixed Models Analysis; Difference in LS mean = 0.025, 95% CI 2-sided [-0.012 to 0.062]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.0038, Mixed Models Analysis; Difference in LS mean = 0.055, 95% CI 2-sided [0.018 to 0.092]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.0241, Mixed Models Analysis; Difference in LS mean = 0.048, 95% CI 2-sided [0.006 to 0.090]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = 0.093, 95% CI 2-sided [0.051 to 0.134]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.0461, Mixed Models Analysis; Difference in LS mean = 0.044, 95% CI 2-sided [0.001 to 0.087]
Statistical Analysis 8: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.0037, Mixed Models Analysis; Difference in LS mean = 0.064, 95% CI 2-sided [0.021 to 0.107]

38. Secondary Outcome: Change From Baseline in EuroQol Quality of Life 5-Dimension 5-Level Scale (EQ-5D-5L)- Visual Analogue Scale Score at Week 2, 4, 8 and 12
Description: EQ-5D-5L is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score. EQ-5D-5L consists of two components: a health state profile and an optional VAS. EQ-5D VAS was used to record a participant's (aged above 17 years) rating for his/her current health-related quality of life state and captured on a vertical VAS (0-100), where 0 = worst imaginable health state and 100 = best imaginable health state.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 121 | 119 | 60
units on a scale
  Change at Week 2 | 5.586 [3.203 to 7.969] | 9.697 [7.294 to 12.100] | 1.038 [-2.361 to 4.437]
  Change at Week 4 | 6.207 [3.473 to 8.940] | 11.931 [9.174 to 14.688] | 1.846 [-2.005 to 5.696]
  Change at Week 8 | 6.982 [3.847 to 10.117] | 10.740 [7.642 to 13.838] | 0.937 [-3.528 to 5.402]
  Change at Week 12 | 8.604 [5.509 to 11.699] | 10.409 [7.328 to 13.489] | -1.035 [-3.451 to 5.520]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0319, Mixed Models Analysis; Difference in LS mean = 4.548, 95% CI 2-sided [0.397 to 8.700]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = 8.659, 95% CI 2-sided [4.496 to 12.822]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.0702, Mixed Models Analysis; Difference in LS mean = 4.361, 95% CI 2-sided [-0.362 to 9.084]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Difference in LS mean = 10.085, 95% CI 2-sided [5.349 to 14.821]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.0300, Mixed Models Analysis; Difference in LS mean = 6.045, 95% CI 2-sided [0.589 to 11.501]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.0005, Mixed Models Analysis; Difference in LS mean = 9.803, 95% CI 2-sided [4.368 to 15.237]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.0067, Mixed Models Analysis; Difference in LS mean = 7.569, 95% CI 2-sided [2.119 to 13.019]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.0008, Mixed Models Analysis; Difference in LS mean = 9.374, 95% CI 2-sided [3.933 to 14.815]

39. Secondary Outcome: Change From Baseline in EuroQol Quality of Life 5-Dimension Youth Scale (EQ-5D-Y): Index Value at Week 2, 4, 8 and 12
Description: EQ-5D-Y: standardized participant (aged 12-17 years) completed questionnaire consisted of 2 components: a health state profile and an optional VAS. EQ-5D health state profile had 5 dimensions: mobility, self-care, usual activities, pain/discomfort, anxiety/depression. Each dimension has 5 levels: 1= no problems, 2= slight problems, 3= moderate problems, 4= severe problems, and 5= extreme problems. Responses to 5 dimensions comprised a health state/a single utility index value. E.g. if a participant responded "no problems" for each 5 dimensions, then health state was coded as "11111" with a predefined index value to it. Every health state (coded as combination of responses on each of 5 dimensions) had a unique predefined utility index value assigned to it, by EuroQol. UK value sets (with all possible health states) was used for adolescents in the study, range from 1 to -0.594. Higher (positive) scores = better health state.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 31 | 32 | 16
units on a scale
  Change at Week 2 | 0.115 [0.039 to 0.191] | 0.209 [0.134 to 0.284] | 0.119 [0.009 to 0.228]
  Change at Week 4 | 0.168 [0.071 to 0.265] | 0.278 [0.183 to 0.374] | -0.006 [-0.149 to 0.137]
  Change at Week 8 | 0.122 [0.017 to 0.228] | 0.198 [0.093 to 0.304] | 0.118 [-0.040 to 0.275]
  Change at Week 12 | 0.160 [0.056 to 0.265] | 0.215 [0.109 to 0.322] | 0.153 [-0.007 to 0.314]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.9568, Mixed Models Analysis; Difference in LS mean = -0.004, 95% CI 2-sided [-0.137 to 0.130]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.1782, Mixed Models Analysis; Difference in LS mean = 0.090, 95% CI 2-sided [-0.042 to 0.223]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.0491, Mixed Models Analysis; Difference in LS mean = 0.174, 95% CI 2-sided [0.001 to 0.347]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.0015, Mixed Models Analysis; Difference in LS mean = 0.284, 95% CI 2-sided [0.112 to 0.456]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.9638, Mixed Models Analysis; Difference in LS mean = 0.004, 95% CI 2-sided [-0.185 to 0.194]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.4016, Mixed Models Analysis; Difference in LS mean = 0.080, 95% CI 2-sided [-0.109 to 0.270]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.9429, Mixed Models Analysis; Difference in LS mean = 0.007, 95% CI 2-sided [-0.184 to 0.198]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.5212, Mixed Models Analysis; Difference in LS mean = 0.062, 95% CI 2-sided [-0.130 to 0.254]

40. Secondary Outcome: Change From Baseline in EuroQol Quality of Life 5-Dimension Youth Scale (EQ-5D-Y): Visual Analogue Scale Score at Week 2, 4, 8 and 12
Description: EQ-5D-Y is a standardized participant completed questionnaire that measures health-related quality of life and translates that score into an index value or utility score specifically developed and validated for use by youths age 12-17 years. EQ-5D-Y consists of two components: a health state profile and an optional VAS. EQ-5D VAS was used to record a participant's rating for his/her current health-related quality of life state and captured on a vertical VAS (0-100), where 0 = worst imaginable health state and 100 = best imaginable health state.
Time Frame: Baseline, Week 2, 4, 8, 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 32 | 32 | 16
units on a scale
  Change at Week 2 | 5.515 [0.318 to 10.712] | 14.933 [9.742 to 20.124] | 3.384 [-4.217 to 10.985]
  Change at Week 4 | 5.359 [-0.339 to 11.057] | 15.496 [9.803 to 21.188] | -1.494 [-10.060 to 7.072]
  Change at Week 8 | 11.828 [5.736 to 17.919] | 12.510 [6.345 to 18.674] | 3.156 [-6.213 to 12.524]
  Change at Week 12 | 10.347 [5.347 to 15.347] | 17.224 [12.151 to 22.297] | 4.276 [-3.397 to 11.948]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.6467, Mixed Models Analysis; Difference in LS mean = 2.131, 95% CI 2-sided [-7.095 to 11.358]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 1]; Test type: Superiority; p = 0.0147, Mixed Models Analysis; Difference in LS mean = 11.549, 95% CI 2-sided [2.338 to 20.761]
Statistical Analysis 3: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.1894, Mixed Models Analysis; Difference in LS mean = 6.853, 95% CI 2-sided [-3.453 to 17.159]
Statistical Analysis 4: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 3]; Test type: Superiority; p = 0.0015, Mixed Models Analysis; Difference in LS mean = 16.990, 95% CI 2-sided [6.699 to 27.281]
Statistical Analysis 5: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.1267, Mixed Models Analysis; Difference in LS mean = 8.672, 95% CI 2-sided [-2.518 to 19.862]
Statistical Analysis 6: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 5]; Test type: Superiority; p = 0.1009, Mixed Models Analysis; Difference in LS mean = 9.354, 95% CI 2-sided [-1.866 to 20.573]
Statistical Analysis 7: Comparison: PF-04965842 100 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.1915, Mixed Models Analysis; Difference in LS mean = 6.071, 95% CI 2-sided [-3.107 to 15.249]
Statistical Analysis 8: Comparison: PF-04965842 200 mg vs Placebo; [analysis description as in outcome 5, analysis 7]; Test type: Superiority; p = 0.0064, Mixed Models Analysis; Difference in LS mean = 12.948, 95% CI 2-sided [3.754 to 22.143]

41. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy Fatigue Scale (FACIT-F) at Week 12
Description: FACIT-F is a 13-item questionnaire. Participants (aged above 17 years) scored each item on a 5-point scale: 0 (not at all) to 4 (very much). Higher the participant's response to the questions (with the exception of 2 negatively stated) greater was the participant's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the FACIT-F score for a total possible score of 0 (worse score) to 52 (the best score) where higher scores indicated better overall health status (less fatigue).
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 106 | 108 | 49
units on a scale | 2.4 [0.8 to 3.9] | 3.3 [1.7 to 4.8] | -1.3 [-3.6 to 1.0]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; Test type: Superiority; p = 0.0102, ANCOVA — Analysis of covariance (ANCOVA) model was used including treatment as main effect and randomization strata (baseline disease severity and age category) and baseline value as covariates; Difference in LS mean = 3.6, 95% CI 2-sided [0.9 to 6.4]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; Test type: Superiority; p = 0.0013, ANCOVA — ANCOVA model was used including treatment as main effect and randomization strata (baseline disease severity and age category) and baseline value as covariates; Difference in LS mean = 4.5, 95% CI 2-sided [1.8 to 7.3]

42. Secondary Outcome: Change From Baseline in Pediatric Functional Assessment of Chronic Illness Therapy Fatigue Scale (Peds-FACIT-F) at Week 12
Description: Peds-FACIT-F is a 13-item questionnaire for adolescents of 12-17 years of age. Participants scored each item on a 5-point scale: 0 (none of the time) to 4 (all of the time). Higher the participant's response to the questions (with the exception of 2 negatively stated), greater was the participant's fatigue. For all questions, except for the 2 negatively stated ones, the code was reversed and a new score was calculated as (4 minus the participant's response). The sum of all responses resulted in the Peds-FACIT-F score for a total possible score of 0 (worse score) to 52 (the best score) where higher scores indicated better overall health status (less fatigue).
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 31 | 30 | 13
units on a scale | 2.2 [0.5 to 3.9] | 2.1 [0.3 to 3.8] | 1.2 [-1.4 to 3.9]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; Test type: Superiority; p = 0.5241, ANCOVA — [p-value comment as in outcome 41, analysis 2]; Difference in LS mean = 1.0, 95% CI 2-sided [-2.1 to 4.2]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; Test type: Superiority; p = 0.5821, ANCOVA — [p-value comment as in outcome 41, analysis 2]; Difference in LS mean = 0.9, 95% CI 2-sided [-2.3 to 4.1]

43. Secondary Outcome: Change From Baseline in Short Form-36v2 (SF-36v2) Acute Summary Score at Week 12: Physical Component Summary
Description: SF-36v2 health survey is a self-administered questionnaire consisting of 36 questions, measuring 8 health domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. These domains were also summarized as physical and mental component summary scores. Physical component summary: the minimum score is 0 and the maximum score is 100. Higher scores indicates a better health state.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 106 | 108 | 50
units on a scale | 4.3 [3.0 to 5.6] | 5.2 [3.9 to 6.5] | 0.5 [-1.4 to 2.4]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; Test type: Superiority; p = 0.0013, ANCOVA — [p-value comment as in outcome 41, analysis 2]; Difference in LS mean = 3.8, 95% CI 2-sided [1.5 to 6.1]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — [p-value comment as in outcome 41, analysis 2]; Difference in LS mean = 4.7, 95% CI 2-sided [2.4 to 7.0]

44. Secondary Outcome: Change From Baseline in Short Form-36v2 Acute Summary Score at Week 12: Mental Component Summary
Description: SF-36v2 health survey is a self-administered questionnaire consisting of 36 questions, measuring 8 health domains: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health. These domains were also summarized as physical and mental component summary scores. Mental component summary: the minimum score is 0 and the maximum score is 100. Higher scores indicates a better health state.
Time Frame: Baseline, Week 12
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
Number analyzed (Participants) | 106 | 108 | 50
units on a scale | 1.5 [-0.1 to 3.0] | 2.8 [1.3 to 4.3] | -0.2 [-2.5 to 2.0]
Statistical Analysis 1: Comparison: PF-04965842 100 mg vs Placebo; Test type: Superiority; p = 0.2256, ANCOVA — [p-value comment as in outcome 41, analysis 2]; Difference in LS mean = 1.7, 95% CI 2-sided [-1.0 to 4.4]
Statistical Analysis 2: Comparison: PF-04965842 200 mg vs Placebo; Test type: Superiority; p = 0.0275, ANCOVA — [p-value comment as in outcome 41, analysis 2]; Difference in LS mean = 3.0, 95% CI 2-sided [0.3 to 5.8]

45. Secondary Outcome: Plasma Concentration Versus Time Summary of PF-04965842
Description: Concentration versus time summary was calculated by setting concentration values below the lower limit of quantification (LLQ) = =1.00 nanogram per milliliter (ng/mL) to zero.
Time Frame: Day 1 of Week 4: 0 hour(Pre-dose), 0.5 hours post-dose; Day 1 of Week 12: 0.5, 4 hours post-dose
Population: Analysis set included all randomized participants who received at least 1 dose of PF-04965842 and had pharmacokinetic measurements. Here, 'Number Analyzed' = participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg
Number analyzed (Participants) | 142 | 144
ng/mL
  Week 4: 0 Hour | 14.57 (65.044) | 58.16 (162.11)
  Week 4: 0.5 Hour post dose: number analyzed (Participants) | 116 | 121
  Week 4: 0.5 Hour post dose | 485.3 (393.36) | 889.7 (786.96)
  Week 12: 0.5 Hour Post-dose: number analyzed (Participants) | 103 | 106
  Week 12: 0.5 Hour Post-dose | 440.6 (373.81) | 933.9 (741.09)
  Week 12: 4 Hour Post-dose: number analyzed (Participants) | 119 | 122
  Week 12: 4 Hour Post-dose | 273.1 (176.37) | 838.9 (544.29)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 16
Description: Same event may appear as adverse event (AE) and serious AE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as nonserious in another participant or 1 participant may have experienced both serious and nonserious event during study.
Arm/Group | PF-04965842 100 mg | PF-04965842 200 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/156 | 0/154 | 0/77
Serious Adverse Events (participants affected / at risk) | 5/156 | 5/154 | 3/77
Other Adverse Events (participants affected / at risk) | 65/156 | 65/154 | 26/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04965842 100 mg (N=156) | PF-04965842 200 mg (N=154) | Placebo (N=77)
Retinal detachment (Eye disorders) | 1 | 0 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 1
Peritonsillitis (Infections and infestations) | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-04965842 100 mg (N=156) | PF-04965842 200 mg (N=154) | Placebo (N=77)
Nausea (Gastrointestinal disorders) | 14 | 31 | 2
Nasopharyngitis (Infections and infestations) | 23 | 18 | 8
Upper respiratory tract infection (Infections and infestations) | 11 | 11 | 5
Headache (Nervous system disorders) | 12 | 15 | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 22 | 8 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT03349060/SAP_000.pdf
  • Study Protocol (2018-06-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT03349060/Prot_001.pdf